CLINICAL TRIAL: NCT07366476
Title: Effectiveness of Electrical Stimulation and Biofeedback on Fecal Incontinence in Children With Repaired Anorectal Malformation: A Comparative Randomized Clinical Trial
Brief Title: Effectiveness of Electrical Stimulation and Biofeedback on Fecal Incontinence in Children With Repaired Anorectal Malformation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Collaborators: El Galaa Teaching Hospital (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, Lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HG000124
Record Dates: First submitted 2025-12-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Fecal Incontinence (FI); Anorectal Malformations
Keywords: fecal incontinence; anorectal malformation; biofeedback; anal electrical stimulation; pelvic floor muscles training
MeSH Terms: conditions — Fecal Incontinence; Anorectal Malformations | interventions — Behavior Therapy; Biofeedback, Psychology; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: randomized comparative clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: who run the randomization process
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): receive anal electrical stimulation, pelvic floor muscles training, and behavioral therapy
  Interventions: Behavioral: behavioral therapy; Device: electrical stimulation; Other: pelvic floor muscles training
- Combined group (Experimental): receive animated biofeedback in combination with anal electrical stimulation and behavioral therapy
  Interventions: Behavioral: behavioral therapy; Device: biofeedback; Device: electrical stimulation

INTERVENTIONS:
Behavioral: behavioral therapy — instructions, diet and toilet modification, motivation and reinforcement
Device: biofeedback — animated biofeedback for pelvic floor muscles training
  Arms: Combined group
Device: electrical stimulation — anal electrical stimulation to stimulate pelvic floor muscles
Other: pelvic floor muscles training — exercises to reeducate pelvic floor muscles control
  Arms: ES group

SUMMARY:
This study aimed to investigate and compare the effect of electrical stimulation and biofeedback with electrical stimulation alone on fecal incontinence in children with repaired imperforate anus, with ages from 6 to 10 years.

DETAILED DESCRIPTION:
A comparative, randomized, clinical trial regarding children who complain of fecal incontinence after operative repair of imperforate anus, to evaluate the effect of biofeedback assisted pelvic floor muscles training through animated games combined with anal electrical stimulation and anal electrical stimulation with pelvic floor muscles training through measuring anal muscles activity and implementing a bowel diary.

ELIGIBILITY:
Inclusion Criteria:

* children with repaired anorectal malformation
* evident spared anal sphincter muscles by MRI
* the age range from 6 to 10 years
* able to follow instructions
* Faecal symptoms will be evaluated for a month to confirm study eligibility.

Exclusion Criteria:

* children with absent anal sphincter muscles by MRI
* children with post-colon surgery other than ARM
* neurologic/neuropathic disorder
* sensory or hearing deficits
* psychological disturbances.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
anal sphincter muscle activity | before and after 3 months of treatment
  The anal sphincter muscles, comprising the internal and external sphincters, play a critical role in maintaining continence and regulating the release of feces. In the context of fecal incontinence in children with repaired anorectal malformation, the activity of these muscles is crucial for understanding their functional restoration post-surgery. Electrical stimulation and biofeedback therapies aim to enhance the tone and coordination of these muscles, improving their ability to control defecation. By assessing the activity of the anal sphincter muscles through method like pressure measurement, the study will determine how these interventions influence muscle function and whether they contribute to a reduction in fecal incontinence episodes. The analysis of sphincter muscle activity is key in evaluating the effectiveness of these therapies in strengthening the muscles and improving overall bowel control.

SECONDARY OUTCOMES:
fecal soiling frequency | a weak before treatment and the last weak of treatment
  Fecal soiling refers to the involuntary leakage of small amounts of stool or mucus, which can result in stains or marks on clothing or bedding. This condition is often associated with fecal incontinence, where individuals are unable to control the release of stool. Fecal soiling frequency refers to how often these incidents occur within a given timeframe, typically measured over a day, week, or month.
  The frequency of fecal soiling can vary significantly from one individual to another, depending on the severity of incontinence, the functionality of the anal sphincters, and other factors such as diet, bowel habits, and the effectiveness of any treatments or interventions. It is often used as a key indicator in clinical studies to assess the effectiveness of treatments for fecal incontinence, such as biofeedback, electrical stimulation, or pelvic floor rehabilitation.
  Tracking fecal soiling frequency helps clinicians understand the patient's condition, determine the severity of their

CONTACTS AND LOCATIONS:
Overall Officials: Rabab S Mohamed, PhD, Principal Investigator — El Galaa Teaching Hospital
Locations (1):
- El-Galaa Teaching Hospital, Cairo, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided